CLINICAL TRIAL: NCT01604980
Title: Use of Indicator Amino Acid Oxidation Technique to Determine Protein Requirement of Elderly Female Subjects >75 Years Old
Brief Title: Determination of Protein Requirements in Elderly Female Subjects >75 Yrs Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Senior Scientist, The Research Institute, Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0019850580-B
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Healthy Females; Protein Requirement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Protein Intakes (Experimental): subjects will recieve differnt levels of protein intakes varying from 0.2 to2.0g/kg/day.
  Interventions: Dietary Supplement: Protein intake.

INTERVENTIONS:
Dietary Supplement: Protein intake. — protein intakes will be varied at 0.2, 0.5, 0.7, 0.9, 1.0, 1.2, 1.5, 1.8 and 2.0g/kg/day

SUMMARY:
Minimal data are available on protein requirements throughout the lifespan. Currently available recommendations are based on nitrogen balance data. The limitations of the nitrogen balance method have been well described. Importantly, nitrogen balanced underestimates requirements.

The current DRI requirement for healthy adult males is based on the reanalysis of the nitrogen balance date from Young and Scrimshaw. This data was reanalyzed statistically by Rand et al. and he concluded that the protein requirement of healthy adults was 0.65 and 0.83 (mean and RDA) g/kg/day of good quality protein. Using IAAO, the investigators group estimated the protein requirement of young men (mean age 27 years) to be 0.93 and 1.2 g/kg/day (mean and RDA).

Currently there are no studies on protein requirement in the elderly. In a recent nutrition survey conducted by NHANES, the authors concluded that adults between the ages of 51 - 70 years old consumed an average on 1.0 g/kg/day (ideal body weight) of protein which represents about 15 % of calories. Depending on the calculations used for ideal body weight some older adults could be getting higher or lower than requirement. There is no scientifically derived protein estimate for older adults. Therefore there is a need to measurer protein requirement in that population.

The goal of this study therefore is to measure the protein requirement of female elderly subjects >75 years using the IAAO technique.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elderly females >75 years
2. Willingness to participate in the study
3. Females without a chronic disease or acute illness that could affect protein and AA metabolism eg, diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
4. Females with hypertension if well controlled by medications -

Exclusion Criteria:

1. Presence of disease known to affect protein and AA requirement and synthesis like diabetes, cancer, liver o kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
2. On medications known to affect protein and amino acid metabolism like e.g. steroids.
3. Significant weight loss during the past month.
4. Individual on weight reducing diets.
5. Inability to tolerate the diet or unwilling to have blood drawn from a venous access for the purposes of the study.
6. Significant coffee consumption of more than 2 cups/day (400 mg of caffeine/day)
7. Significant Alcohol consumption of more than one drink/day ( 1 beer, ½ glass of wine) -

Ages: 76 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
13CO2 Production | Study Day 3
  Urine and breath samples will be collected on day 3 of the experiment to determine the rate of production

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rafii M, Chapman K, Owens J, Elango R, Campbell WW, Ball RO, Pencharz PB, Courtney-Martin G. Dietary protein requirement of female adults >65 years determined by the indicator amino acid oxidation technique is higher than current recommendations. J Nutr. 2015 Jan;145(1):18-24. doi: 10.3945/jn.114.197517. Epub 2014 Oct 15. PMID 25320185